CLINICAL TRIAL: NCT06440447
Title: EXploring Patterns of Use and Effects of Adult Day Programs to Improve Trajectories of Continuing CarE (EXPEDITE)
Brief Title: EXploring Patterns of Use and Effects of Adult Day Programs to Improve Trajectories of Continuing CarE
Acronym: EXPEDITE
Status: Not yet recruiting | Type: Observational
Sponsor: York University (Other)
Collaborators: Carswell Family Foundation (Unknown); Alzheimer Society of York Region (Unknown)
Responsible Party: Principal Investigator, Matthias Hoben, Associate Professor, Helen Carswell Chair in Dementia Care, York University
Other Study IDs: 563198b
Record Dates: First submitted 2024-05-16; First posted 2024-06-03 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Adult Day Programs; Continuing Care; Old Age; Dementia; Family/friend Caregivers
Keywords: Adult day programs; Older adults; Program evaluation; Cohort studies; Health administrative data
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Day program attendees: Older adults (65+ years) attending an adult day program in Alberta, British Columbia, or Manitoba
  Interventions: Other: Adult day program use
- Non-attendees: Older adults with an initial Resident Assessment Instrument - Home Care (RAI-HC), who are not attending a day program in Alberta, British Columbia, or Manitoba
  Interventions: Other: Other community care (non-attendees)

INTERVENTIONS:
Other: Adult day program use — Day program use patterns will be determined, using Latent Class Analysis. Three continuous variables will be categorized as low, low-moderate, high-moderate, high, using sample distribution quartiles: (1) Time between first RAI-HC assessment and first attendance of a day program, (2) average number of hours of day program attendance (i.e., total number of hours spent in a day program divided by the number of times attended), and (3) total number of days a person attended a day program.
  Groups: Day program attendees
Other: Other community care (non-attendees) — Any publicly funded continuing care services in the community, other than adult day programming (e.g., home care, in-home respite). Community care participants will be propensity score matched with day program participants, using RAI-HC variables on day program eligibility (to ensure similarity of non-attendees to day program attendees). Matching variables will include: physical functioning, cognition, behavioural symptoms, bladder/bowel continence, availability of a caregiver, and caregiver distress. The investigators will also include variables on health and social characteristics (e.g., age, sex, type/duration of publicly funded community care received before the matching index date, deprivation indices).
  Groups: Non-attendees

SUMMARY:
This study seeks to understand the impact of Canada's adult day program on attendees and non-attendees, especially those with dementia and other co-morbidities. A retrospective cohort study will be conducted, including older adults in the community who do or do not attend adult day programs in Alberta, British Columbia, and Manitoba, Canada. The objectives are to (1) compare patterns of day program use (including non-use) by Canadian province (Alberta, British Columbia, Manitoba), and time, (2) compare characteristics of older adults by day program use pattern (including non-use), province, and time, and (3) to examine whether those who are exposed to day programs, compared to a propensity-score matched comparison group of non-exposed older adults in the community, enter long-term care homes at later times (primary outcome), are less likely to have depressive symptoms, physical and cognitive change, and have lower use of primary, acute, and emergency care (secondary outcomes).

DETAILED DESCRIPTION:
Adult day programs provide critical supports to both, older adults living in the community, and their family/friend caregivers. This is essential because ensuring high-quality care in the community for as long as possible and avoiding or delaying long-term care home admissions are key priorities of older adults, their caregivers, and healthcare systems. While most older adults in Canada receive care in the community, about 10% of newly admitted nursing home residents have relatively low care needs that could be met in the community with the right supports. Caregivers provide most of the care in the community, which puts them at high risk for caregiver burden. Day programs intend to mitigate these issues by providing respite to caregivers. However, research on the effectiveness of day programs is inconsistent. Generally, the methodological quality of studies is poor, and especially Canadian research is lacking. The research objectives are to (1) explore changes in patterns of day program use (including non-use) between provinces and over time, (2) compare characteristics of older adults with different day program use patterns (including non-use), and (3) assess whether day program attendees compared to a propensity score matched control group of non-attendees have better outcomes. This retrospective cohort study will use population-based clinical and health administrative data of older adults (65+ years) who received publicly subsidized continuing care in the community in Alberta, British Columbia, and Manitoba between January 01, 2012 and December 31, 2024. Patterns of day program use (i.e., variations in time to attend a day program for the first time, and frequency and duration of attendance) and how these patterns vary by province and over time will be assessed. Characteristics of older adults with different patterns of day program use (e.g., no, low, medium, high) will be compared. Characteristics of the participants will include age, sex, dementia status, frailty level, comorbidity status, socioeconomic status, availability of a caregiver, and caregiver distress. Finally, propensity-matched comparison group (by region, age, gender, cognitive/physical impairment, type/duration of community care received previously) of older adults who have not attended a day program will be created. Time-to-event models and general estimating equations will assess whether day program attendees compared to non-attendees enter continuing care facilities later (primary outcome); use emergency, acute, or primary care less frequently; experience less cognitive and physical decline; and have better mental health (secondary outcomes). Models will include day program exposure as an independent variable and will be adjusted for province, participant demographics, medical and functional conditions, caregiver availability/distress, other community services received (e.g., home care, in-home respite), and (if appropriate) matching variables.

ELIGIBILITY:
Inclusion criteria:

* Persons aged 65 years and over
* Initial RAI-HC assessment completed
* Attendance of an adult day program (for cohort 1)
* Receipt of any community-based continuing care services, other than adult day program (cohort 2)

Exclusion criteria:

- No receipt of any community-based continuing care service

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study focuses on community care systems in Alberta, British Columbia, and Manitoba, all of which assess day program eligibility using comparable processes, criteria, and assessments (i.e. RAI-HC). The yearly average number of completed RAI-HC assessments is ~20,000-30,000 in Alberta, ~34,000-39,000 in British Columbia, and ~10,000 in Manitoba. The estimated number of day program attendees is >20,000/year (>200,000 within the study period), each with multiple assessments.
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to admission to a long-term care homes | From date of home care admission until the date of admission to a long-term care home or loss to follow up (i.e., death, move out of province), whichever came first, assessed up to 12 years (between Jan 31, 2012 and Dec 31, 2024)
  Data will come from provincial continuing care registries, which document the start date of any publicly funded continuing care service a person receives, the end date of this service, and the type of service. The outcome will be the time between a person's first RAI-HC assessment and admission to a long-term care home (i.e., an assisted living home or nursing home).

SECONDARY OUTCOMES:
Symptoms of depression | Baseline (date of home care admission) and annually until study end (Dec 31, 2024) or loss to follow up, whichever came first
  To determine the presence or absence of depressive symptoms, the validated RAI-HC Depression Rating Scale (DRS) will be used. DRS scores range from 0-14, and a cut-point of 3 or higher represents clinically meaningful depressive symptoms.
Presence or absence of physical decline | Baseline (date of home care admission) and annually until study end (Dec 31, 2024) or loss to follow up, whichever came first
  Change in physical functioning will be captured, using the validated RAI-HC Activities of Daily Living Hierarchy (ADLh) scale. The scale ranges from 0 (no impairment) to 6 (maximum impairment), and the outcome will be dichotomous, indicating any increase (versus no change or a decrease) between the previous and follow up measurement in this scale.
Presence or absence of cognitive decline | Baseline (date of home care admission) and annually until study end (Dec 31, 2024) or loss to follow up, whichever came first
  Change in cognition will be captured, using the validated RAI-HC Cognitive Performance Scale (CPS). The scale ranges from 0 (no impairment) to 6 (maximum impairment), and the outcome will be dichotomous, indicating any increase (versus no change or a decrease) between the previous and follow up measurement in this scale.
Emergency room registrations | Baseline (date of home care admission) and annually until study end (Dec 31, 2024) or loss to follow up, whichever came first
  The National Ambulatory Care Report System (NACRS) captures all emergency department visits and diagnoses. The outcome will be the yearly average number of a person's emergency department visits.
Hospital stays | Baseline (date of home care admission) and annually until study end (Dec 31, 2024) or loss to follow up, whichever came first
  The Discharge Abstract Database (DAD) includes information on all inpatient hospital stays, including diagnoses and length of stay. The outcome will be the yearly average number of a person's hospital stays.
Primary care provider visits | Baseline (date of home care admission) and annually until study end (Dec 31, 2024) or loss to follow up, whichever came first
  Care provider claims data includes health service claims submitted for payment by primary care providers (e.g., general practitioners, nurse practitioners, geriatricians, geriatric psychiatrists, neurologists, therapists). The outcome will be the yearly average number of a person's primary care provider visits.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Hoben, PhD, Principal Investigator — York University

IPD SHARING:
Plan to Share IPD: No
The health administrative data used in this study are owned by the respective provincial health authorities. Provincial data policies do not allow public sharing of these data. The research team will work with an in-house health system data analyst in each of the provinces to carry out the analyses. Data are required to stay within the respective province and within the province's protected and secure data repository.

REFERENCES:
- [Background] European Commission. The 2018 ageing report: Economic and budgetary projections for the 28 EU member states (2016-2070). Luxembourg: European Commission; 2018. Report No.: 79. Available from: https://economy-finance.ec.europa.eu/publications/2018-ageing-report-economic-and-budgetary-projections-eu-member-states-2016-2070_en#files [accessed Sep 2, 2022]
- [Background] Federal/provincial/territorial ministers responsible for seniors. Core community supports to age in community. Ottawa: Government of Canada; 2019. Available from: https://www.canada.ca/en/employment-social-development/corporate/seniors/forum/core-community-supports.html [accessed Sep 2, 2022]
- [Background] MacDonald B-J, Wolfson M, Hirdes JP. The future co$t of long-term care in Canada. Toronto, ON: National Institute on Aging; 2019. Available from: https://www.nia-ryerson.ca/reports [accessed Sep 2, 2022]
- [Background] Thomas KS, Applebaum R. Long-term services and supports (LTSS): A growing challenge for an aging America. Public Policy & Aging Report 2015;25(2):56-62. doi: 10.1093/ppar/prv003
- [Background] Whitman DB. Unsolved mysteries in aging policy. Public Policy & Aging Report 2015;25(2):67-73. doi: 10.1093/ppar/prv006
- [Background] 2022 Alzheimer's disease facts and figures. Alzheimers Dement. 2022 Apr;18(4):700-789. doi: 10.1002/alz.12638. Epub 2022 Mar 14. PMID 35289055
- [Background] Prince MJ, Wimo A, Guerchet MM, Ali GC, Wu Y-T, Prina M. World Alzheimer Report 2015 - The Global Impact of Dementia: An analysis of prevalence, incidence, cost and trends. London: Alzheimer's Disease International; 2015. Available from: https://www.alzint.org/resource/world-alzheimer-report-2015/ [accessed Sep 2, 2022
- [Background] Public Health Agency of Canada. Dementia in Canada. Ottawa: Public Health Agency of Canada; Available from: https://www.canada.ca/en/public-health/services/publications/diseases-conditions/dementia.html [accessed Sep 2, 2022]
- [Background] Nguyen H, Manolova G, Daskalopoulou C, Vitoratou S, Prince M, Prina AM. Prevalence of multimorbidity in community settings: A systematic review and meta-analysis of observational studies. J Comorb. 2019 Aug 22;9:2235042X19870934. doi: 10.1177/2235042X19870934. eCollection 2019 Jan-Dec. PMID 31489279
- [Background] The Academy of Medical Sciences. Multimorbidity: a priority for global health research. London: The Academy of Medical Sciences; 2018. Available from: https://acmedsci.ac.uk/policy/policy-projects/multimorbidity [accessed Sep 2, 2022]
- [Background] Canadian Institute for Health Information (CIHI). Quick stats - Home Care Reporting System (HCRS) profile of clients in home care 2020-2021. Available from: https://www.cihi.ca/en/quick-stats [accessed Sep 2, 2022]
- [Background] Morgan T, Ann Williams L, Trussardi G, Gott M. Gender and family caregiving at the end-of-life in the context of old age: A systematic review. Palliat Med. 2016 Jul;30(7):616-24. doi: 10.1177/0269216315625857. Epub 2016 Jan 26. PMID 26814213
- [Background] Quesnel-Vallée A, Willson A, Reiter-Campeau S. Health inequalities among older adults in developed countries: Reconciling theories and policy approaches. In: George L, Ferraro K, editors. Handbook of aging - social sciences 8th ed. London: Elsevier; 2016.
- [Background] Quesnel-Vallée A, Farrah J-S, Jenkins T. Population aging, health systems, and equity: Shared challenges for the United States and Canada. In: Settersten Jr. RA, Angel JL, editors. Handbook of sociology of aging New York, Dordrecht, Heidelberg, London: Springer; 2011.
- [Background] McGrail K. Long-term care as part of the continuum. Healthc Pap. 2011;10(4):39-43; discussion 58-62. doi: 10.12927/hcpap.2011.22190. PMID 21593615
- [Background] Sinha S, Dunning J, Wong I, Nicin M, Nauth S. Enabling the future provision of long-term care in Canada. Toronto, ON: National Institute on Aging; 2019. Available from: https://www.nia-ryerson.ca/reports [accessed Sep 2, 2022]
- [Background] Federal/provincial/territorial ministers responsible for seniors. Report on housing needs of seniors. Ottawa: Government of Canada; 2019. Available from: https://www.canada.ca/en/employment-social-development/corporate/seniors/forum/report-seniors-housing-needs.html [accessed Sep 2, 2022]
- [Background] Spasova S, Baeten R, Coster S, Ghailani D, Peña-Casas R, Vanhercke art. Challenges in long-term care in Europe - A study of national policies 2018. Brussels: European Commission; 2018. Available from: https://ec.europa.eu/social/main.jsp?langId=en&catId=1135&newsId=9185&furtherNews=yes [accessed Sep 2, 2022]
- [Background] Goncalves J, Weaver F, Konetzka RT. Measuring State Medicaid Home Care Participation and Intensity Using Latent Variables. J Appl Gerontol. 2020 Jul;39(7):731-744. doi: 10.1177/0733464818786396. Epub 2018 Jul 6. PMID 29978735
- [Background] Wysocki A, Butler M, Kane RL, Kane RA, Shippee T, Sainfort F. Long-Term Services and Supports for Older Adults: A Review of Home and Community-Based Services Versus Institutional Care. J Aging Soc Policy. 2015;27(3):255-79. doi: 10.1080/08959420.2015.1024545. PMID 25942005
- [Background] Royal Bank of Canada. 2013 RBC retirement myths & realities poll: most appealing living arrangements for boomers. 2013. Available from: http://www.rbc.com/newsroom/news/2013/20131024-myths-realities.html [accessed Sep 2, 2022]
- [Background] American Association of Retired Persons (AARP). 2018 home and community preferences: A national survey of adults age 18-plus. Washington, DC: AARP Research; 2018. Available from: https://www.aarp.org/research/topics/community/info-2018/2018-home-community-preference.html [accessed Sep 2, 2022]
- [Background] European Commission. Health and long-term care in the European Union. Luxembourg: European Commission; 2007. Available from: https://sid-inico.usal.es/idocs/F8/FDO22761/health_european_union.pdf [accessed Sep 2, 2022]
- [Background] Gutman GM, Milstein S, Killam J, Lewis D, Hollander MJ. Adult Day Care centres in British Columbia: models, characteristics and services. Health Rep. 1993;5(2):189-207. English, French. PMID 8292758
- [Background] Gutman GM, Milstein S, Killam J, Lewis D, Hollander MJ. Adult day care centres in British Columbia: client characteristics, reasons for referral and reasons for non-attendance. Health Rep. 1993;5(3):321-33. English, French. PMID 8199334
- [Derived] Hoben M, Maxwell CJ, Ubell A, Doupe MB, Goodarzi Z, Allana S, Beleno R, Berta W, Bethell J, Daly T, Ginsburg L, Rahman AS, Nguyen H, Tate K, McGrail K. EXploring Patterns of Use and Effects of Adult Day Programs to Improve Trajectories of Continuing Care (EXPEDITE): Protocol for a Retrospective Cohort Study. JMIR Res Protoc. 2024 Aug 30;13:e60896. doi: 10.2196/60896. PMID 39213024